CLINICAL TRIAL: NCT00971607
Title: Sevoflurane Sedation During Primary Percutaneous Coronary Intervention.
Brief Title: Sevoflurane In Acute Myocardial Infarction
Acronym: SIAMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shahar Lavi, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-09-165; 15793 (Other: REB)
Record Dates: First submitted 2009-07-09; First posted 2009-09-03 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Postconditioning; Sevoflurane
MeSH Terms: interventions — Oxygen; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Sevoflurane
  Interventions: Drug: Oxygen + Sevoflurane
- 2 (Placebo Comparator): Oxygen
  Interventions: Drug: Oxygen (placebo)

INTERVENTIONS:
Drug: Oxygen + Sevoflurane — Oxygen with end-tidal MAC of Sevoflurane 0.5 during PCI.
  Arms: 1
Drug: Oxygen (placebo) — Control will receive oxygen only.
  Arms: 2

SUMMARY:
Ischemic postconditioning can reduce myocardial injury following myocardial infarction.

A potential pharmacological agent is the anesthetic Sevoflurane. The investigators' hypothesis is that sevoflurane during primary percutaneous coronary intervention (PCI) will reduce infarct size.

DETAILED DESCRIPTION:
Patients with first STEMI that will be treated by primary PCI, will be randomized to sedation with Sevoflurane during the procedure or to usual care.

ELIGIBILITY:
Inclusion Criteria:

* First STEMI, presenting within 6 hours after the onset of chest pain
* Symptoms lasting > 30 minutes
* Persistent ST-segment elevation > 0.1 mV in 2 or more contiguous leads

Exclusion Criteria:

* Hypersensitivity to sevoflurane or other halogenated agents
* Malignant hyperthermia
* Cardiac arrest
* Cardiogenic shock
* Previous myocardial infarction or coronary bypass surgery
* Pre-infarction angina
* Heart failure (NYHA III/IV)
* Chronic inflammatory disease
* Severe renal impairment
* Hepatic dysfunction
* Use of Glyburide

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Infarct size by area under the curve of cardiac markers. | 3 days

SECONDARY OUTCOMES:
Left ventricular function. | Six month
ST segment elevation resolution | 90 minutes
TIMI flow | 60 minutes
Renal function | 48 hours
CRP | 24 hours
Patient satisfaction | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Lavi, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sceinces Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Lavi S, Alemayehu M, McCarty D, Warrington J, Lavi R. One-year outcome of the sevoflurane in acute myocardial infarction randomized trial. Can J Anaesth. 2015 Dec;62(12):1279-86. doi: 10.1007/s12630-015-0456-2. Epub 2015 Aug 22. PMID 26296299